CLINICAL TRIAL: NCT05278689
Title: Jejunal Feeding Via Gastrojejunal Tube in Refractory Gastroesophageal Reflux
Acronym: ReJej
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP-ReJej
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastrojejunal; Children; GERD (Gastroesophageal reflux disease)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Gastroesophageal reflux disease (GERD) in children can be severe and lead to multiple complications, dizziness, esophagitis, respiratory failure or ENT infections.

In the case of resistance to treatment with proton pump inhibitors (PPIs), alternatives treatments includes antireflux surgery or fasting associated with parenteral nutrition. The use of gastrointestinal tubes (GJT) is relatively recent. Its objective is to allow a direct jejunal feeding, thus limiting the risk of severe gastroesophageal reflux disease (GERD). Jejunal feeding using GJT has been compared to surgical techniques without finding any superiority. However, the risk of GERD recurrence appears to be greater if anti-reflux surgery is performed in a young child. As an alternative to anti-reflux surgery, prolonged parenteral nutrition (NPE) is burdened with its own morbidity (metabolic, infectious, vascular). In addition, the natural course of GERD is usually towards spontaneous improvement with the age and growth of the child. GJT may be used to postpone anti-reflux surgery and prevent NPE while waiting for spontaneous GERD improvement. In a cohort of 27 children, 5 did not require surgery or parenteral nutrition after placement of GJT . However, this study is difficult to analyze because of 9/27 deaths. Complications from GJT are common, ranging from obstruction requiring replacement to jejunal perforation. We will study the benefit of jejunal feeding on YSG for children followed for severe GERD.

References :

1. Srivastava R, Downey EC, O'Gorman M, Feola P, Samore M, Holubkov R, et al. Impact of fundoplication versus gastrojejunal feeding tubes on mortality and in preventing aspiration pneumonia in young children with neurologic impairment who have gastroesophageal reflux disease. Pediatrics 2009; 123:338-45.
2. Stone B, Hester G, Jackson D, Richardson T, Hall M, Gouripeddi R, et al. Effectiveness of Fundoplication or Gastrojejunal Feeding in Children With Neurologic Impairment. Hosp Pediatr 2017; 7:140-8.
3. Michaud L, Coopman S, Guimber D, Sfeir R, Turck D, Gottrand F. Percutaneous gastrojejunostomy in children: efficacy and safety. Arch Dis Child 2012; 97:733-4.
4. Campwala I, Perrone E, Yanni G, Shah M, Gollin G. Complications of gastrojejunal feeding tubes in children. J Surg Res 2015; 199:67-71.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) in children can be severe and lead to multiple complications, among them dizziness, esophagitis, respiratory failure or ENT infections. In the case of resistance o proton pump inhibitors (PPIs) therapy, alternatives treatments includes anti-reflux surgery or fasting associated with parenteral nutrition.

The use of gastrointestinal tubes (GJT) is relatively recent. Its objective is to allow a direct jejunal feeding, thus limiting the risk of severe gastroesophageal reflux disease (GERD).

Jejunal feeding using GJT has been compared to surgical techniques without finding any superiority.

However, the risk of GERD recurrence appears to be greater if anti-reflux surgery is performed at a young age.

As an alternative to anti-reflux surgery, prolonged parenteral nutrition (PN) is burdened with its own morbidity (metabolic, infectious, vascular).

In addition, the natural course of GERD is usually towards spontaneous improvement with the age and growth of the child. GJT may be used to postpone anti-reflux surgery and prevent PN while waiting for spontaneous GERD improvement.

Literature data found in a cohort of 27 children, 5 did not require surgery or parenteral nutrition after placement of GJT. However, this study is difficult to analyze because of 9/27 deaths.

Complications from GJT are common, ranging from obstruction of the tube requiring replacement to jejunal perforation that is a life treating condition.

This monocentric, retrospective study will be conducted at a French pediatric university hospital. The study was approved by hospital's ethics committee and aims to help to evaluate the potential advantages of GJT feeding in hospital settings among patients admitted with severe GERD and determine if this feeding route may prevent or postpone recourse to invasive procedures like surgery or alternative nonsurgical treatments like parenteral nutrition (PN) that have morbidity in order to control the reflux disease and its complications and at the same time prevent growth deficit among affected children.

The data will be entered on an e-CRF (Epidata) from the patient files consulted on site by the investigators or a person delegated by them. The data will be anonymized when entered with only the order number, initials and year of birth of the patients. The correspondence table will be kept in each participating center by the local investigator. Only professionals involved in this study will have access to the pseudonymised database. Data will be recorded on a restricted access server. Persons with direct access to the data take all necessary precautions to ensure the confidentiality of this data. The anonymized data will be stored on secure servers not connected to the Internet.

The quantitative variables will be described in mean and standard deviation. Qualitative variables will be described in numbers (percent). Comparison tests. Qualitative data will be analyzed with Chi2 or Fischer's exact test. The qualitative values will be analyzed using Student's t-test if their distribution is normal or by the non-parametric Mann-Whitney test. Multivariate analysis will use logistic regression to study age, weight and initial pathology. The significance threshold was set at p < 0.05

The primary outcomes are :

Need for invasive GERD treatments, anti-reflux surgery or parenteral nutrition 1 month after Gastrojejunal tube placement and at the end of follow-up.

Secondary outcomes are:

Duration of use of Gastrojejunal tube. type of the Gastrojejunal tube

The following criteria will be compared before and after the installation of Gastrojejunal tube :

* Anti-reflux treatments
* Complications of GERD: respiratory, dizziness
* Duration of hospitalization
* Intussusception, Dumping syndrome,
* Mechanical complications: obstruction, extrajejunal displacement, extraction, rupture of the GJT
* Weight and height

References :

1. Srivastava R, Downey EC, O'Gorman M, Feola P, Samore M, Holubkov R, et al. Impact of fundoplication versus gastrojejunal feeding tubes on mortality and in preventing aspiration pneumonia in young children with neurologic impairment who have gastroesophageal reflux disease. Pediatrics 2009; 123:338-45.
2. Stone B, Hester G, Jackson D, Richardson T, Hall M, Gouripeddi R, et al. Effectiveness of Fundoplication or Gastrojejunal Feeding in Children With Neurologic Impairment. Hosp Pediatr 2017; 7:140-8.
3. Michaud L, Coopman S, Guimber D, Sfeir R, Turck D, Gottrand F. Percutaneous gastrojejunostomy in children: efficacy and safety. Arch Dis Child 2012; 97:733-4.
4. Campwala I, Perrone E, Yanni G, Shah M, Gollin G. Complications of gastrojejunal feeding tubes in children. J Surg Res 2015; 199:67-71.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18
* Insertion of a gastro-jejunal tube with a goal of feeding by the jejunal route during GERD beyond 1/1/2000
* Follow-up> 4 months.
* Follow-up at Robert-Debré hospital

Exclusion Criteria:

* Refusal to participate in the study
* intra-gastric Gastro-jejunal tube placement, with the aim of gastric emptying

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hospitalized patients with more than 4 months follow-up
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-11-19 (Estimated); Study Completion 2022-11-19 (Estimated)

PRIMARY OUTCOMES:
GERD "Gastroesophageal Reflux Disease" treatments | 4 months
  Need for invasive GERD treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital - Assistance Publique Hopitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Faccioli N, Sierra A, Mosca A, Bellaiche M, Lengline H, Bonnard A, Viala J. Jejunal Feeding by Gastrojejunal Tube in Pediatric Refractory Gastroesophageal Reflux Disease. J Pediatr Gastroenterol Nutr. 2023 Aug 1;77(2):267-273. doi: 10.1097/MPG.0000000000003785. Epub 2023 Mar 31. PMID 37477887